CLINICAL TRIAL: NCT07065214
Title: Argon Plasma Treatment for Ovarian Endometrioma Compared to Standard Cystectomy: A Prospective Controlled Randomized Pilot Study
Brief Title: Argon Plasma Treatment for Ovarian Endometrioma Compared to Standard Cystectomy
Acronym: OVAPLAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erbe Elektromedizin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OVAPLAS
Record Dates: First submitted 2025-06-12; First posted 2025-07-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis
Keywords: ovarian endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard cystectomy (Other): Investigator uses lap bipolar forceps for endometrioma treatment (standard treatment)
  Interventions: Device: Lap bipolar forceps
- APC treatment (Experimental): Investigator uses APC applicator for endometrioma treatment. This is a CE approved device
  Interventions: Device: APC

INTERVENTIONS:
Device: APC — For the surgical procedure for ovarian endometrioma treatment APCapplicator will be used
  Other Names: APC Treatment with APCapplicator
  Arms: APC treatment
Device: Lap bipolar forceps — For ovarian endometrioma treatment the standard of care treatment will be performed.
  Arms: Standard cystectomy

SUMMARY:
The study is a prospective, monocentric, randomized controlled, two-armed, pilot-study conducted at Department for Women's Health, Tuebingen, Germany.

In this Post Market Study it will be determined whether and to what extent the two surgical procedures for ovarian endometrioma treatment (standard cystectomy versus APC) may affect the ovarian reserve by comparing changes in serum AMH levels after treatment.

Seventy-two (72) patients who meet all eligibility criteria will undergo surgical procedure. The patients will be randomized into the group with standard cystectomy treatment or with APC treatment. Per group n=36 patients will be treated i.e., 1:1 randomization.

A pre-specified primary endpoint analysis is planned after the last patient has undergo Visit 4 (Follow-up after 6 months) to analyze the primary endpoint.

Screening takes place during the first visit (V1). During the second visit (V2) the participants will receive the ovarian endometriosis treatment procedure either with the APC or the standard cystectomy. Standard procedure (standard cystectomy) will be performed for additional endometriosis lesions. The follow up visits (V3 - V5) will take place after three, six and twelve months. Visit 3 and Visit 4 will take place at the study site and AMH will be measured. Whereas Visit 5 will take place via telemedical contact, i.e. phone call.

ELIGIBILITY:
Inclusion Criteria:

* Indication for surgical endometrioma treatment according to patient symptoms
* Signed informed consent

Exclusion Criteria:

* Expected lack of patient compliance or inability of the patient to understand the purpose of the clinical trial
* Prior procedures at the ovaries
* Recurrent endometrioma (patients with recurrent endometriosis outside of the ovar, e.g. peritoneal endometriosis lesions can be included)
* Pregnant or breastfeeding patients
* Participation in any other clinical study that could affect the AMH level or pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of AMH (Anti-Müller hormone) level | Screening Visit 1 (up to -28 days before day 0); Visit 3 (day 0 +3 months +/- 14 days; Visit 4 (day 0 + 6 months +/- 14 days)
  The comparison of patient AMH changes (ΔAMH) before and after surgery (Follow up Visit after 3 and 6 months) with either APC or standard cystectomy (ΔAMH Group 1 versus ΔAMH Group 2).

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Krämer, Prof. Dr. med., Principal Investigator — Department for Women's Health, Tuebingen, Germany
Locations (1):
- Department for Women's Health, Tübingen, Germany, Germany

REFERENCES:
- [Background] Younis JS, Shapso N, Ben-Sira Y, Nelson SM, Izhaki I. Endometrioma surgery-a systematic review and meta-analysis of the effect on antral follicle count and anti-Mullerian hormone. Am J Obstet Gynecol. 2022 Jan;226(1):33-51.e7. doi: 10.1016/j.ajog.2021.06.102. Epub 2021 Jul 13. PMID 34265271
- [Background] Stefanovic S, Sutterlin M, Gaiser T, Scharff C, Neumann M, Berger L, Froemmel N, Tuschy B, Berlit S. Microscopic, Macroscopic and Thermal Impact of Argon Plasma, Diode Laser, and Electrocoagulation on Ovarian Tissue. In Vivo. 2023 Mar-Apr;37(2):531-538. doi: 10.21873/invivo.13111. PMID 36881055
- [Background] Lockyer EK, Schreurs A, Lier M, Dekker J, Melgers I, Mijatovic V. Treatment of ovarian endometriomas using plasma energy in endometriosis surgery: effect on pelvic pain, return to work, pregnancy and cyst recurrence. Facts Views Vis Obgyn. 2019 Mar;11(1):49-55. PMID 31695857
- [Background] Working group of ESGE, ESHRE, and WES; Saridogan E, Becker CM, Feki A, Grimbizis GF, Hummelshoj L, Keckstein J, Nisolle M, Tanos V, Ulrich UA, Vermeulen N, De Wilde RL. Recommendations for the surgical treatment of endometriosis-part 1: ovarian endometrioma. Gynecol Surg. 2017;14(1):27. doi: 10.1186/s10397-017-1029-x. Epub 2017 Dec 19. PMID 29285022
- [Background] Muzii L, Achilli C, Bergamini V, Candiani M, Garavaglia E, Lazzeri L, Lecce F, Maiorana A, Maneschi F, Marana R, Perandini A, Porpora MG, Seracchioli R, Spagnolo E, Vignali M, Benedetti Panici P. Comparison between the stripping technique and the combined excisional/ablative technique for the treatment of bilateral ovarian endometriomas: a multicentre RCT. Hum Reprod. 2016 Feb;31(2):339-44. doi: 10.1093/humrep/dev313. Epub 2015 Dec 18. PMID 26682578